CLINICAL TRIAL: NCT05988866
Title: Effects of a Digital Health Application (Lipodia) on LDL-cholesterol Levels in Individuals With LDL-cholesterol Levels Above Recommended Targets for Reducing Cardiovascular Risk: Randomized Controlled Trial
Brief Title: Effects of a Digital Health Application (Lipodia) on LDL-cholesterol Levels
Acronym: DIGICHOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University of Kiel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: lipodia RCT 2025
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Hypercholesterolemia; Dyslipidemias
Keywords: LDL-C; digital intervention
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants allocated to the intervention group will receive access to lipodia in addition to treatment as usual (TAU).
  lipodia is a digital health application designed for individuals with hypercholesterinemia, accessible through a web browser. The application focuses on treatment methods derived health behavior change and cognitive behavioral therapy (CBT). Topics addressed by lipodia are activity planning and impulse control, dietary habits, physical activity, stress management, mood management, sleep management, weight management, as well as quitting smoking and drinking.
  The program operates through interactive "dialogues", which are accompanied by illustrations, audio recordings, motivating text messages, worksheets, and summaries. Users are also encouraged to regularly complete short questionnaires to monitor their complaints. Once registered, the program remains accessible for 365 days.
  Interventions: Behavioral: lipodia
- Control group (No Intervention): Participants allocated to the control group will receive access to treatment as usual (TAU).

INTERVENTIONS:
Behavioral: lipodia — Participants will receive access to the digital health intervention lipodia in addition to TAU.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to find out if lipodia, a digital health intervention, can help lower cholesterol levels and improve other health measures in adults with high cholesterol.

The main questions it aims to answer are:

* Does lipodia, together with regular treatment, lower LDL cholesterol (bad cholesterol) better than regular treatment alone?
* Does lipodia help improve other health outcomes, like how confident participants feel in managing their health?

Researchers will compare two groups:

* Intervention group: Participants use the lipodia intervention and continue their usual treatment.
* Control group: Participants continue with their usual treatment only.

Participants will:

* Fill out questionnaires online and visit a certified lab at the start of the study, after 3 months, and after 6 months
* Have blood tests at each lab visit to check their cholesterol and other blood fat levels
* Continue with their usual treatment (both groups) and use lipodia, a digital health app, for six months (intervention group only)

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18
* Diagnosis of hypercholesterolemia (ICD-10 E78.0, E78.2, E78.4, E78.5, E78.8, E78.9) confirmed by a laboratory test and physician diagnosis
* LDL-C levels above risk-adapted target
* TG levels < 400 mg/dL
* Stability of potential drug treatment during the last 4 weeks
* Stability of potential hormonal treatment during the last 6 months
* Patient was made aware of lifestyle measures by GP or specialist
* Consent to participation
* Sufficient knowledge of the German language

Exclusion criteria

* Homozygous Familial Hypercholesterolemia (FH), given that it is a genetic condition which is relatively unresponsive to lifestyle changes
* Hyperlipidemia type III, given that it is a genetic condition which is relatively unresponsive to lifestyle changes
* Patients receiving plasmapheresis
* Lp(a) > 50 mg/dL
* current pregnancy or planned pregnancy during the study period
* planned major operations
* liver dysfunction
* end-stage renal failure
* other systemic conditions that might interfere with successful study participation
* Plans to change drug (including hormonal) treatment in the upcoming 6 months
* Use of another digital intervention for hypercholesterolemia/dyslipidemia in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fasting LDL-C levels | 6 months

SECONDARY OUTCOMES:
Patients' activation | 6 months
  Assessed with the total score of the PAM-13. Higher scores indicate higher patient activation (better outcome).
Fasting non-HDL-C levels | 6 months
Health-related quality of life | 6 months
  Assessed with the total score of the AQoL-8D. Higher scores indicate higher quality of life (better outcome).
BMI | 6 months
Fasting triglyceride levels | 6 months
Fasting HDL-C levels | 6 months
Fasting LDL-C levels | 3 months

OTHER OUTCOMES:
Patients' activation | 3 months
  Assessed with the total score of the PAM-13. Higher scores indicate higher patient activation (better outcome).
Fasting non-HDL-C levels | 3 months
Health-related quality of life | 3 months
  Assessed with the total score of the AQoL-8D. Higher scores indicate higher quality of life (better outcome).
BMI | 3 months
Fasting triglyceride levels | 3 months
Fasting HDL-C levels | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Jauch-Chara, Prof., Principal Investigator — Christian-Albrechts-Universität zu Kiel
Locations (1):
- GAIA AG, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No